CLINICAL TRIAL: NCT01540799
Title: Pathway M-1: Sphenopalatine Ganglion Stimulation for the AcuteTreatment of High Disability Migraine Headache
Acronym: Pathway M-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pathway M-1 (CIP-003)
Record Dates: First submitted 2012-02-20; First posted 2012-02-29 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2017-05

CONDITIONS: High Frequency, High Disability Migraine
Keywords: Migraine; High disability migraine; Sphenopalatine ganglion; Neuromodulation; Neurostimulation; Autonomic nervous system
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: ATI Neurostimulation System
- Other (Other): Stimulation not able to be felt
  Interventions: Device: ATI Neurostimulation System

INTERVENTIONS:
Device: ATI Neurostimulation System — ATI Neurostimulator (NS-100) and Remote Controller (RC-200)

SUMMARY:
The purpose of the clinical study is to evaluate the use of an implanted sphenopalatine ganglion (SPG) neurostimulator for the treatment of migraine headache pain, migraine headache symptoms and migraine frequency in high disability migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Subject has been diagnosed at least 3 months prior to study enrollment with migraine headache with or without aura according to the 2004 ICHD-II criteria 1.1 or 1.2.1.1.
* Subject reports at least 75% of migraine attacks having predominantly fixed (non side-shifting) unilateral temporal or ocular pain.
* Subject reports that moderate/severe migraine pain is typically preceded by a mild pain phase.
* Subject reports a minimum of 8 days per month and a maximum of 14 days per month with migraine attacks of at least moderate severity based on the subject/Investigator's knowledge for at least 3 months prior to inclusion and confirmed for at least 1 month during the Pre-Implant Baseline Period using the Pathway M-1 Daily Headache Diary.
* Subject reports at least 24 hours of pain-free periods between typical migraine attacks.
* Subject has a MIDAS grade of III or IV, or has a HIT-6 score > 56.
* Subject is medically intractable in the opinion of the Investigator.
* Subject has had stable type and dosage of preventive headache medications for at least 1 month prior to study enrollment and agrees to maintain stable type and dosage of preventive headache medications through the completion of the Experimental Period.
* Subject is able to distinguish migraine attacks from other headaches (i.e., TTH).
* Subject agrees to not participate in supplemental or alternative therapy through the Open Label phase of the study. This includes: acupuncture, spinal manipulation, TENS, and magnetic fields treatments.
* Subject has the ability to read, comprehend, and to reliably record information as required by the Protocol.
* Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Subject's overall health, age and/or comorbidities place subject at high risk for complications from surgery and/or general anesthesia.
* Subject has been diagnosed with chronic migraine during the last year according to 2006 ICHD-IIR Appendix 1.5.1.
* Subject currently has Medication Overuse Headache (MOH) or has a history of MOH during the last year according to the ICHD-2R 2006 criteria.
* Subject has used any triptans, pain medications or analgesics of any kind for any indication on more than 14 days per month over the last three months.
* Subject reports continuous daily headaches for one month or longer at time of consent.
* Subject reports initial onset of migraines within the last year.
* Subject has undergone facial surgery or has metallic implants in the area of the pterygopalatine fossa or zygomaticomaxillary buttress ipsilateral to the planned implant site that, in the opinion of the Investigator, may lead to the inability to properly implant or use the Neurostimulator.
* Subject has active oral or dental abscess.
* Subject has been treated with therapeutic radiation to the facial region.
* Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past 6 months or require periodic MRI follow-up.
* Subject's pterygomaxillary fissure is less than 1.2 mm in width at the level of the vidian canal, as determined by CT scan.
* Subject has clinically significant drug (including opioid) or alcohol abuse as defined by DSM-IV-TR, will likely be unable to refrain from substance abuse throughout the study, has other significant pain problem, substance abuse or active depressive episode that might confound the study assessments in the opinion of the Investigator.
* Subject is currently participating or has participated in the last month in another clinical study in which the subject has, is, or will be exposed to an investigational drug or device.
* Subject is felt to be at risk of non-compliance (e.g., for completing the diary, maintaining a stable headache medicine regimen or returning for required follow-up visits) in the Investigator's opinion.
* Subject is a woman of childbearing age who is pregnant, nursing, or not using contraception. A sterilized or infertile woman is exempt from the requirement to use contraception.
* Subject has had previous lesional radiofrequency ablation of the ipsilateral sphenopalatine ganglion (SPG).
* Subject has had blocks or non-lesional pulsed RF of the ipsilateral SPG in the last 3 months.
* Subject has undergone botulinium toxin injections of the head and/or neck in the last 3 months.
* Subject has or requires a pacemaker/defibrillator or other implantable device having a sense amplifier that is programmed 'On.'
* Subject has a history of bleeding disorders or coagulopathy or is unable to discontinue anticoagulation, antiplatelet, or GP IIb IIIa inhibitor medication in preparation for the implantation procedure.
* Subject has a chronic neurological illness of the face (e.g., facial nerve paralysis, trigeminal neuralgia).
* Subject is not suitable for the study for any reason in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Major Device- and Surgical-Related Complications | Implantation through completion of Experimental Period (18 weeks following the implantation procedure)
  Occurrence rate of death, any surgery or hospitalization due to deterioration in subject health, or other Major Device-related Adverse Events
Effective Therapy | During Experimental Period (12 to 18 weeks following implantation)
  Number of Migraine Pain Days during the Experimental Period, compared between the Treatment and Control arms.
  Migraine Pain Day is any calendar day that:
  1. Has less than 4 hours of moderate or severe pain meeting criteria C and D for migraine ICHD-II 1.1 AND
  2. No Acute Headache or Migraine Pain Medication (pharmacologic medications, not including SPG stimulation, used to treat acute headache pain).
     AND
  3. No SPG stimulation is applied for headache pain of any intensity

OTHER OUTCOMES:
Number of Migraine Free Days during the Experimental Period, compared between the Treatment and Control arms. | During Experimental Period (12 to 18 weeks following implantation)
  Migraine Free Day is any calendar day that:
  1. Has less than 4 hours of moderate or severe pain meeting criteria C and D for migraine ICHD-II 1.1 AND
  2. No Acute Headache or Migraine Pain Medication is used AND
  3. No SPG stimulation is applied for headache pain of any intensity
Number of Headache Free Days during the Experimental Period, compared between the Treatment and Control arms | During Experimental Period (12 to 18 weeks following implantation)
  Headache Free Day is any calendar day that:
  1. Has less than 4 hours of moderate or severe pain AND
  2. No Acute Headache or Migraine Pain Medication is used AND
  3. No SPG stimulation is applied for headache pain of any intensity
Percent change in number of Migraine Free Days during the last 4 weeks of the Experimental Period relative to the 4 weeks preceding the implantation procedure, compared between the Treatment and Control arms | During Experimental Period (14 to 18 weeks following implantation) compared to Baseline
Percent change in number of Headache Free Days during the last 4 weeks of the Experimental Period relative to the 4 weeks preceding the implantation procedure, compared between the Treatment and Control arms | During Experimental Period (14 to 18 weeks following implantation) compared to Baseline
Descriptive responder analysis of Migraine Free Days during the Experimental Period relative to the Pre-Implant Baseline | During Experimental Period (12 to 18 weeks following implantation) compared to Baseline
Descriptive responder analysis of Headache Free Days during the Experimental Period relative to the Pre-Implant Baseline | During Experimental Period (12 to 18 weeks following implantation) compared to Baseline
Proportion of subjects who achieve Pain Relief at 4 hours in at least 50% of their moderate/severe SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Proportion of subjects who achieve Pain Relief at 2 hours in at least 50% of their moderate/severe SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Proportion of subjects who achieve Pain Freedom at 4 hours in at least 50% of their moderate/severe SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Proportion of subjects who achieve Pain Freedom at 2 hours in at least 50% of their moderate/severe SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Proportion of subjects who achieve Pain Freedom at 4 hours in at least 50% of their mild SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Proportion of subjects who achieve Pain Freedom at 2 hours in at least 50% of their mild SPG stimulation treated attacks during the Experimental Period | During Experimental Period (12 to 18 weeks following implantation)
Descriptive analysis of associated symptoms [i.e., photophobia, phonophobia, nausea/vomiting, autonomic symptoms] relief at 4 hours, evaluated for relief of each symptom individually and for relief of all symptoms | During Experimental Period (12 to 18 weeks following implantation)
Disability and Quality of Life as categorized by the HIT-6, MIDAS and SF-36v2 surveys administered at the end of the Experimental Period, compared between the Treatment and Control arms | End of Experimental Period (18 weeks following implantation)
Descriptive responder analysis of Disability and Quality of Life as categorized by the HIT-6, MIDAS and SF-36v2 surveys relative to the Pre-Implant Baseline survey responses | End of Experimental Period (18 weeks following implantation) compared to Baseline
Global patient evaluation of SPG stimulation therapy (very poor, poor, no opinion, good, very good) administered at the end of the Experimental Period, compared between the Treatment and Control arms | End of Experimental Period (18 weeks following implantation)
Use of preventive medications during the Open Label Period as compared to Baseline, evaluated in all subjects | During Open Label Period (18 to 52 weeks following implantation) compared to Baseline
Use of acute medications during the Experimental Period as compared between the Treatment and Control arms | During Experimental Period (12 to 18 weeks following implantation)
Use of acute medications during the Open Label Period as compared to Baseline, evaluated in all subjects | During Open Label Period (18 to 52 weeks following implantation) compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor Jensen, MD, PhD, Principal Investigator — Danish Headache Center, Glostrup Hospital
Locations (3):
- Dept. of Neurology, K12 Bldg. 1st fl, De Pintelaan 185 B-9000, Ghent, Belgium
- Danish Headache Center & Department of Neurology, Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Copenhagen, Denmark
- Servicio de Neurologia, Hospital Clinico Universitario, Valencia, Spain